CLINICAL TRIAL: NCT02408445
Title: Body Composition in Infants With Klinefelter Syndrome and Effects of Testosterone Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-1720; UL1TR001082 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Klinefelter Syndrome
Keywords: body composition; Klinefelter syndrome; XXY; sex chromosome variation; sex chromsome aneuploidy
MeSH Terms: conditions — Klinefelter Syndrome | interventions — testosterone 17 beta-cypionate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone treatment (Experimental): Testosterone cypionate (200 mg/ml) intramuscular injection
  Interventions: Drug: testosterone cypionate 200mg/ml
- No treatment (No Intervention): Subjects will not receive any testosterone during the study period.

INTERVENTIONS:
Drug: testosterone cypionate 200mg/ml — Subjects in this group will be randomized to receive testosterone cypionate 200 mg/ml to be given intramuscularly every 4 weeks for a total of 3 doses.
  Arms: Testosterone treatment

SUMMARY:
This research study in infant males with Klinefelter syndrome (47,XXY) will learn more about body composition (muscle and fat) and male hormones and look at the effect of testosterone shots on body composition. The Investigators know that older boys and men with Klinefelter syndrome often have more fat compared to muscle than adults without Klinefelter syndrome, but we do not know if this difference is present at birth or develops over time. The Investigators will learn if body composition and motor skills are improved with testosterone treatment in infants with Klinefelter syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male infants with 47,XXY karyotype

Exclusion Criteria:

* Gestational age at birth <36 weeks
* Birth weight <5%ile or >95% for gestational age
* History of thrombosis in a first degree relative
* Exposure to androgen therapy outside of the study protocol.

Ages: 42 Days to 108 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanlee M Davis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone Treatment | No Treatment
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Treatment | No Treatment | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: days] | 73 (22) | 70 (23) | 72 (22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 9 | 17
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Fat Percent Z-score
Description: Body fat percentage will be measured using air displacement plethysmography (PEA POD) at the beginning and end of the study period. Age and sex-normed z-scores will be calculated. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean with negative numbers indicating values lower than the mean and positive values higher. Change in the z-score over time, if following a normal growth curve, is 0. Positive change in z-scores indicates a gain in body fat above growth typically expected. Negative change in z-scores indicates a gain in body fat that is less than typically expected.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
score on a scale | -0.12 (0.65) | 0.92 (0.62)

2. Secondary Outcome: Serum Luteinizing Hormone (LH)
Description: Serum will be collected at the first study visit prior to randomization. Ultrasensitive LH will be measured.
Time Frame: baseline only
Population: Analysis was completed only on subjects for which sufficient blood was able to be obtained and that has been measured at this time.
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 6 | 8
mIU/mL | 2.5 (1.1) | 2.5 (1.3)

3. Secondary Outcome: Serum Follicle Stimulating Hormone (FSH)
Description: Serum will be collected at the first study visit prior to randomization. Ultrasensitive FSH will be measured.
Time Frame: baseline only
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 6 | 8
mIU/mL | 1.8 (0.3) | 1.7 (0.5)

4. Secondary Outcome: Serum Total Testosterone
Description: Serum will be collected at the first study visit prior to randomization. Total testosterone by mass spectroscopy will be measured.
Time Frame: baseline only
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 6 | 8
ng/dl | 181 (100) | 166 (30)

5. Secondary Outcome: Serum Inhibin B (INHB)
Description: Serum will be collected at the first study visit prior to randomization. Inhibin B levels will be measured.
Time Frame: baseline only
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 8 | 6
pg/ml | 244 (96) | 355 (151)

6. Secondary Outcome: Serum Anti-Mullerian Hormone (AMH)
Description: Serum will be collected at the first study visit prior to randomization. AMH levels will be measured.
Time Frame: baseline only
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 6 | 8
pmol/l | 1377 (688) | 2208 (862)

7. Secondary Outcome: Leptin
Description: Serum will be collected at the first study visit prior to randomization. Leptin levels will be measured.
Time Frame: baseline only
Population: Unable to be analyzed due to insufficient quantities of serum collected. Prioritized hormone assays first.
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Raw Score on the Alberta Infant Motor Scale
Description: Muscle tone and motor development will be assessed by an occupational therapist using the standardized Alberta Infant Motor Scale (AIMS). The AIMS scale measures infant motor maturation from birth until the age of independent walking. An occupational therapists assesses 58 motor behavior items in 4 position categories: prone (21 items), supine (9 items), sitting (12 items) & standing(16 standing). Each item receives one point (range of raw scores 0-58), with higher scores indicating more skills acquired. For change in scores, the raw score at 3 months was subtracted from the baseline raw score.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: raw score
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
raw score | 10.5 (4.9) | 8.9 (7.1)

9. Secondary Outcome: Change in Score on the Movement Assessment of Infants (MAI)
Description: Muscle tone and motor development will be assessed by an occupational therapist using the standardized Movement Assessment of Infants (MAI). The MAI evaluates four domains: muscle tone, primitive reflex, automatic reactions and volitional movement. All items are scored 1-5 and summed to generate a "Total Risk Score". Lower scores indicate better function, and Total Risk Scores of 8 or more indicate high risk.
Time Frame: 3 months
Population: Data for this measurement was not collected for any of the participants.
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Total Motor Standard Score on the Peabody Developmental Motor Scales 2
Description: Motor development will be assessed by an occupational therapist using the standardized Peabody Developmental Motor Scales 2. Standard scores are normalized to age with a mean of 100 and standard deviation of 15. Change in standard score was calculated as the differences between the subject's standard score at 3 months minus the standard score at baseline. A positive change in standard scores would indicate greater growth on the measure relative to peers, while a negative number would indicate slower growth on the measure relative to peers.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: change in standard score
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
change in standard score | 2.8 (7.3) | 2.0 (6.9)

11. Secondary Outcome: Change in Penile Length
Description: Stretched penile length will be measured by a physician before randomization and at the end of the study period.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
cm | 0.9 (0.5) | -0.3 (0.6)

12. Secondary Outcome: Change in Fat Free Mass
Description: Fat free mass (lean mass) will be measured using air displacement plethysmography (PEA POD) at the beginning and end of the study period.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Testosterone Treatment | No Treatment
Number analyzed (Participants) | 10 | 10
kg | 1.4 (0.4) | 0.6 (0.3)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse events were captured by parental report in the active treatment arm only. All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed for the 'No Treatment' Arm/Group
Arm/Group | Testosterone Treatment
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Testosterone Treatment (N=10)
Acne (Skin and subcutaneous tissue disorders) | 2 — any parent-reported pimples
Change in diet or elimination habits (Gastrointestinal disorders) | 2 — Parent reported change in appetite, diarrhea, constipation, or other GI-symptom
Erections (Reproductive system and breast disorders) | 3 — Parent report of penile erections (>1 erection noted)
Mood change (General disorders) | 1 — Parent-reported change in mood/demeanor, including irritability, level of alertness, sleepiness, etc.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT02408445/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT02408445/ICF_001.pdf